CLINICAL TRIAL: NCT03543111
Title: Promoting the Psychological Health of Women With SCI: A Virtual World Intervention
Acronym: Zest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency); TIRR Memorial Hermann (Other); University of Montana (Other); Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Susan Robinson-Whelen, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSC-MS-17-0474; H133G080042-10 (Other Grant/Funding Number: National Institute on Disability, Independent Living, and Rehabilitation Research (NIDILRR))
Record Dates: First submitted 2018-05-14; First posted 2018-06-01 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zest (Experimental): Zest is an internet-based psychological health enhancement program for women with spinal cord injury. The intervention will occur in Second Life (SL), which is an online virtual word simulator with a group of women with spinal cord injury.The Zest program will consist of 10 weekly 2-hour group sessions with approximately 8 women using avatars to represent themselves.
  Interventions: Behavioral: Zest
- Control (No Intervention): No intervention - Control participants are provided intervention materials at the end of the study.

INTERVENTIONS:
Behavioral: Zest — Zest is an internet-based psychological health enhancement program for women with spinal cord injury. The intervention will occur in Second Life (SL), which is an online virtual word simulator with a group of women with spinal cord injury.The Zest program will consist of 10 weekly 2-hour group sessions with approximately 8 women using avatars to represent themselves.
  Arms: Zest

SUMMARY:
The purpose of this project is to test the efficacy of an internet-based psychological health enhancement program for women with spinal cord injury. The intervention will occur in Second Life (SL), which is an online virtual word simulator with a group of women with spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* have a traumatic spinal cord injury
* be at least one year post injury
* be able to speak and read English (to participate in the group intervention and complete study questionnaires in English).
* have access to a phone, an email account, and a computer and high-speed Internet connection that meets minimum SL computing requirements.

Exclusion Criteria:

* have a cognitive impairment that significantly limits their ability to give informed consent, participate in the intervention, or complete study assessments as determined by an inability to correctly answer questions on a comprehension of consent questionnaire
* have a significant visual or hearing impairment that would prohibit their ability to participate in the virtual intervention
* report active suicidality
* live in institutions. Individuals living in community-based group and adult foster homes will be invited to participate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must self-identify as a woman during the screening interview.
Enrollment: 175 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Self-esteem as assessed by the Rosenberg Self-Esteem Scale | Baseline
  The effect of the Zest intervention on self-esteem as assessed by the Rosenberg Self-Esteem Scale. This is a 10-item scale with scores ranging from 10-40 with higher scores indicating higher self-esteem.
Self-esteem as assessed by the Rosenberg Self-Esteem Scale | 10 weeks
  The effect of the Zest intervention on self-esteem as assessed by the Rosenberg Self-Esteem Scale. This is a 10-item scale with scores ranging from 10-40 with higher scores indicating higher self-esteem.
Self-esteem as assessed by the Rosenberg Self-Esteem Scale | 6 months
  The effect of the Zest intervention on self-esteem as assessed by the Rosenberg Self-Esteem Scale. This is a 10-item scale with scores ranging from 10-40 with higher scores indicating higher self-esteem.
Depression as assessed by the Patient Health Questionnaire-9 (PHQ-9) | Baseline
  The effect of the Zest intervention on depression as assessed by the Patient Health Questionnaire-9 (PHQ-9). This is a 9-item scale with scores ranging from 0-27 with higher scores indicating more severe depression.
Depression as assessed by the Patient Health Questionnaire-9 (PHQ-9) | 10 weeks
  The effect of the Zest intervention on depression as assessed by the Patient Health Questionnaire-9 (PHQ-9). This is a 9-item scale with scores ranging from 0-27 with higher scores indicating more severe depression.
Depression as assessed by the Patient Health Questionnaire-9 (PHQ-9) | 6 months
  The effect of the Zest intervention on depression as assessed by the Patient Health Questionnaire-9 (PHQ-9). This is a 9-item scale with scores ranging from 0-27 with higher scores indicating more severe depression.
Life satisfaction as assessed by the Satisfaction with Life Scale | Baseline
  The effect of the Zest intervention on life satisfaction as assessed by the Satisfaction with Life Scale. This is a 5-item scale with scores ranging from 5-35 with higher scores indicating greater satisfaction with life.
Life satisfaction as assessed by the Satisfaction with Life Scale | 10 weeks
  The effect of the Zest intervention on life satisfaction as assessed by the Satisfaction with Life Scale. This is a 5-item scale with scores ranging from 5-35 with higher scores indicating greater satisfaction with life.
Life satisfaction as assessed by the Satisfaction with Life Scale | 6 months
  The effect of the Zest intervention on life satisfaction as assessed by the Satisfaction with Life Scale. This is a 5-item scale with scores ranging from 5-35 with higher scores indicating greater satisfaction with life.

SECONDARY OUTCOMES:
Self-efficacy as assessed by the Generalized Self-Efficacy Scale | Baseline
  The effect of the Zest intervention on self-efficacy as assessed by the Generalized Self-Efficacy Scale. This is a 10-item scale with scores ranging from 10-40 with higher scores indicating higher self-efficacy.
Self-efficacy as assessed by the Generalized Self-Efficacy Scale | 10 weeks
  The effect of the Zest intervention on self-efficacy as assessed by the Generalized Self-Efficacy Scale. This is a 10-item scale with scores ranging from 10-40 with higher scores indicating higher self-efficacy.
Self-efficacy as assessed by the Generalized Self-Efficacy Scale | 6 months
  The effect of the Zest intervention on self-efficacy as assessed by the Generalized Self-Efficacy Scale. This is a 10-item scale with scores ranging from 10-40 with higher scores indicating higher self-efficacy.
Social connectedness as assessed by the Medical Outcomes Study Social Support Scale, Emotional/Informational Support subscale. | Baseline
  The effect of the Zest intervention on social connectedness as assessed by the Medical Outcomes Study Social Support Scale, Emotional/Informational subscale. This is an 8-item scale in which scores for each item are averaged. Scores are converted to a 0-100 scale with higher scores indicating more support and, therefore, social connectedness.
Social connectedness as assessed by the Medical Outcomes Study Social Support Scale, Emotional/Informational Support subscale. | 10 weeks
  The effect of the Zest intervention on social connectedness as assessed by the Medical Outcomes Study Social Support Scale, Emotional/Informational subscale. This is an 8-item scale in which scores for each item are averaged. Scores are converted to a 0-100 scale with higher scores indicating more support and, therefore, social connectedness.
Social connectedness as assessed by the Medical Outcomes Study Social Support Scale, Emotional/Informational Support subscale. | 6 months
  The effect of the Zest intervention on social connectedness as assessed by the Medical Outcomes Study Social Support Scale, Emotional/Informational subscale. This is an 8-item scale in which scores for each item are averaged. Scores are converted to a 0-100 scale with higher scores indicating more support and, therefore, social connectedness.
Perceived stress as assessed the by Perceived Stress Scale | Baseline
  The effect of the Zest intervention on perceived stress as assessed by the Perceived Stress Scale. This is a 10-item scale with scores ranging from 0-40 with higher scores indicating more perceived stress.
Perceived stress as assessed the by Perceived Stress Scale | 10 weeks
  The effect of the Zest intervention on perceived stress as assessed by the Perceived Stress Scale. This is a 10-item scale with scores ranging from 0-40 with higher scores indicating more perceived stress.
Perceived stress as assessed the by Perceived Stress Scale | 6 months
  The effect of the Zest intervention on perceived stress as assessed by the Perceived Stress Scale. This is a 10-item scale with scores ranging from 0-40 with higher scores indicating more perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Robinson-Whelen, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (4):
- United States (4):
  - University of Montana, Missoula, Montana
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - TIRR Memorial Hermann, Houston, Texas

REFERENCES:
- [Derived] Robinson-Whelen S, Hughes RB, Gonzalez D, Norah-Davis L, Leon-Novelo LG, Ngan E, Whelen ML, Wenzel L, Taylor HB. Promoting psychological health in women with spinal cord injury: A randomized trial. Rehabil Psychol. 2025 Nov;70(4):426-436. doi: 10.1037/rep0000602. Epub 2025 Feb 6. PMID 39913478

DOCUMENTS (1):
  • Informed Consent Form (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/11/NCT03543111/ICF_000.pdf